CLINICAL TRIAL: NCT00002311
Title: A Phase I-II Dose Escalation Study to Examine the Safety of Four Doses of Wobenzym in HIV Seropositive Patients
Brief Title: The Safety of Four Different Dose Levels of Wobenzym in HIV-Positive Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mucos Pharma GmbH and Co (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 122A
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1993-05

CONDITIONS: HIV Infections
Keywords: Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Wobenzym; Hydrolases
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Wobenzym

INTERVENTIONS:
Drug: Wobenzym

SUMMARY:
To study the safety and efficacy of four different doses of Wobenzym (an enzyme combination consisting of pancreatin, papain, bromelain, trypsin, lipase, amylase, chymotrypsin, and rutin) in patients with HIV infection whose CD4 count is between 250 and 400 cells/mm3. To evaluate the effect of Wobenzym on certain surrogate markers associated with progression of HIV disease.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

HIV seropositivity with CD4 counts between 250 and 400 cells/mm3.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Known hypersensitivity to hydrolytic enzymes such as Wobenzym.
* Known sensitivity to lactose.
* Presumption that the patient will not comply with the dosing schedule or follow-up appointments.

Concurrent Medication:

Excluded:

* Concurrent use of immunosuppressive therapy or steroids.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Saint Luke's - Roosevelt Hosp Ctr, New York, New York, United States